CLINICAL TRIAL: NCT05970367
Title: Impact of an Intensive Motor Rehabilitation Programme Integrating Technology for Adults With Central Neurological Disease: A Randomised Controlled Rehabilitation Study in the Chronic Phase
Brief Title: Intensive Motor Rehabilitation With Technology for Patients With Central Neurological Disease
Acronym: INTeRAcT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: AZ Herentals (Unknown); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Prof., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S67164
Record Dates: First submitted 2023-06-23; First posted 2023-08-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Spinal Cord Injuries; Chronic Disease
Keywords: rehabilitation; intensive; technology
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive rehabilitation program (Experimental): 3 weeks of intensive rehabilitation --> follow-up 9 months standard care
  Interventions: Other: Intensive rehabilitation programme
- Standard care (No Intervention): Follow-up 9 months standard care --> 3 weeks of intensive rehabilitation

INTERVENTIONS:
Other: Intensive rehabilitation programme — Intensive rehabilitation using advanced technology, based on the patient's goals.
  Including cardiovascular fitness training, goal-oriented training, physiotherapy with and without advanced technology and self-management.
  Arms: Intensive rehabilitation program

SUMMARY:
This project will consist of 1 large clinical trial with 3 core concepts: (1) Clinical benefits of an intensive rehabilitation programme using advanced technology, compared to the control group; (2) A full health economic evaluation combined with model-based estimation of costs and benefits; (3) process evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures;
2. A diagnosis of central neurological disease, made by a specialist. Conditions may include stroke or spinal cord injury:

   1. Stroke: Participants must have received a diagnosis of stroke for the first time, have been diagnosed at least 3 months ago, and live at home.
   2. SCI: Participants have a rating A, B, C or D on the American Spinal Injury Association (ASIA) measurement scale, which refers to patients with complete or incomplete impairment. All levels of SCI can be included, if there is a clear patient need linked to the upper and/or lower extremities.
3. At least 3 months post discharge from hospital/rehabilitation centre, living at home;
4. Having a maximum recovery of 85% of independence in daily functioning (FIM/SCIM);
5. Had a normal functional state prior to the pathology: a pre-pathology Barthel Index > 85/100;
6. Unilateral or bilateral weakness of the affected upper or lower limbs (No maximum score in all affected limbs = motricity index: score 5 on 3/3 segments)
7. Having the clinical opportunity to engage in exercise therapy with available technology, assessed by a specialist;
8. Age of > 18 years;
9. Sufficient cognitive ability to understand the games and give informed consent, assessed by a specialist;.

Exclusion Criteria:

1. Having other neurological or musculoskeletal conditions that may affect the protocol, assessed by a specialist;
2. No ability to initiate movements against gravity in the upper and lower limbs;
3. Severe visual impairment, communication, cognitive and language formation problems that would prevent the intervention and measurement process, assessed by a specialist;
4. Any disorder, which in the investigator's opinion might the compromise participant's safety or compliance with the CIP;
5. Female who is pregnant, breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in Functional Independence Measure (FIM) | Baseline - 3weeks - 9months
  The Functional Independence Measure (FIM), which measures independence in daily functioning after stroke. The FIM consists of 18 items designed to assess to what extent a person needs assistance in performing activities of daily living safely and efficiently. The activities consist of a number of basic skills related to self-care, pelvic floor function, transfers, gait, communication and social abilities. The FIM has acceptable reliability and has been found valid in people with stroke.
  Min: 13; Max: 91; Higher = better
Change in Spinal Cord Independence Measure (SCIM) | Baseline - 3weeks - 9months
  Spinal Cord Independence Measure (SCIM), an assessment of achievements of daily function of patients with spinal cord lesions. The scale consists of 19 tasks organized in 3 subscales: self-care, respiration and sphincter management, and mobility. The SCIM is valid and reliable.
  Min: 0; Max: 100; Higher = better

SECONDARY OUTCOMES:
Change in The Canadian Occupational Performance Measure (COPM) | Baseline - 3weeks - 9months
  The Canadian Occupational Performance Measure (COPM), is an evidence-based outcome measure designed to capture a patient's self-perception of performance in everyday living, over time. This outcome can be used in both study populations.
  Min: 1; Max: 10; Higher = better
Change in EQ-5D-5L | Baseline - 3weeks - every month during follow-up - 9 months
  EQ-5D-5L, measures quality of life at five levels of health (mobility, self-care, daily activities, pain/discomfort and anxiety/depression). From this, a weighted health index can be calculated for an individual or population. This scale can also be used for both populations.
  Min: 1; Max: 100; Higher = better
Change in Goal Attainment Scaling (GAS) | Baseline - 3weeks - 9months
  Goal Attainment Scaling (GAS), is an individualised evaluation method. It is scored on an ordinal 5-point scale, which captures a person's individual treatment goal and is scored afterwards on the achievement of that treatment goal. The GAS can and will be used for both stroke and spinal cord injury.
  Min: -2; Max: +2; Higher = better
Change in The fatigue severity scale (FSS) | Baseline - 3weeks - 9months
  The fatigue severity scale (FSS) contains 9 questions assessing the perceived severity of fatigue symptoms in the past week in various daily situations. The patient indicates the extent to which fatigue determines functioning. Again, this will be used for both stroke and spinal cord injury.
  Min: 9; Max: 63; Higher = worse
Borg Rating of Perceived Exertion Scale | During intervention (up to 9 months)
  During the intervention the Borg Rating of Perceived Exertion Scale will be completed to after every therapy block to assess subjective experiences of the patients during physical load.
  Min: 6; Max: 20; Higher = worse
Change in the 6-minute Walk-Test (6MWT) | Baseline - 3weeks - 9months (stroke only)
  The 6-minute Walk-Test (6MWT) is used to measure functional capacity. The maximum distance the patient can cover within 6 minutes is measured.
Change in the action research Arm Test (ARAT) | Baseline - 3weeks - 9months (stroke only)
  The action research Arm Test (ARAT) is an observational measure to assess upper extremity performance (coordination, dexterity and functioning), including 19 items. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally).
  Min: 0; Max: 57; Higher = better
Change in rhe Fugl-Meyer Assessment (FMA) | Baseline - 3weeks - 9months (stroke only)
  The Fugl-Meyer Assessment (FMA) is designed to assess motor functioning in upper and lower limbs, in patients with post-stroke. Patients are assessed on 50 test items and on an ordinal 3-point scale.
  Min: 0; Max: 100; Higher = better
Change in the functional Ambulation Classification (FAC) | Baseline - 3weeks - 9months (stroke only)
  The functional Ambulation Classification (FAC): is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient needs when walking, whether or not they use a personal assistive device.
  Min: 0; Max: 5; Higher = better
Change in the 10 Meter Walk Test (10MWT) | Baseline - 3weeks - 9months (stroke only)
  The 10 Meter Walk Test (10MWT) measures the time needed for a person to walk 10 meters. It is used to determine functional mobility and gait.
Change in the Stroke Self-efficacy Questionnaire | Baseline - 3weeks - 9months (stroke only)
  The Stroke Self-efficacy Questionnaire Evaluate individuals' confidence in carrying out activities of daily living.
  Min: 0; Max: 60; Higher = better

OTHER OUTCOMES:
Change in health economic evaluation | Baseline - 3weeks - every month during follow-up - 9 months
  Through this questionnaire, health economic data are surveyed to estimate direct and indirect costs that participants have due to their condition.
  The following types of resource use will be collected: primary care, emergency visits, inpatient stays, outpatient services, medication, transport costs, the estimation of the amount of informal care, days away from work, and social benefits (e.g. sickness leave payments).
Therapy diary | every month during follow-up (up to 9 months)
  Using a therapy diary that the investigators ask patients to fill in every time they have been to the physical therapist/psychologist. On a monthly basis, these records are requested via mail.
Process evaluation | Structured therapy diaries: during intervention; Semi-structured interviews: 2-4 weeks post intervention; Observations: during intervention
  Structured therapy diaries will document how the intervention is delivered, including session duration and the content of the of exercises.
  Semi-structured interviews with patients and therapists will assess therapy quality, perceived benefits, relevance, satisfaction, and barriers to implementation, as well as expectations for sustainability. Therapists will reflect on adaptations made.
  Observations will deepen understanding of content and delivery: 14 participants will be observed during sessions using a structured scheme. Each therapy type (upper/lower limb, with/without technology, cardiovascular fitness, goal-oriented training, self-management) will be observed weekly over 3 weeks, totaling 6-7 hours per participant per week. Observations will help interpret outcome variations across settings.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Herentals, Herentals
  - KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No